CLINICAL TRIAL: NCT03488537
Title: Detection of Colorectal Cancer From Exhaled Air. Part II: Validation
Brief Title: e-Nose and Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: e-Nose and colorectal cancer
Record Dates: First submitted 2018-03-21; First posted 2018-04-05 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2018-02

CONDITIONS: Colorectal Cancer; Polyps
MeSH Terms: conditions — Colorectal Neoplasms; Polyps

STUDY DESIGN:
Intervention Model Description: This is a Multi center prospective cohort study in subjects eligible for colonoscopy with suspicion for malignant or premalignant lesions of the colon.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients referred for colonoscopy (Other): All patients referred for colonoscopy where invited to participate in our study.
  Interventions: Device: AeonoseTM

INTERVENTIONS:
Device: AeonoseTM — Breath test

SUMMARY:
Colorectal cancer (CRC) is the third most common new cancer diagnosis and a major cause of morbidity and mortality throughout the world. Early detection and treatment are critical factors in the course and prognosis of CRC, and screening programs have proven to be an important means to reduce both CRC related mortality and secondary economic burden.

The diagnostic accuracy of non-invasive screening tests is still limited and a follow-up colonoscopy is required for confirmation of the diagnosis. The faecal occult blood test (FIT) is the most commonly used fecal screening test worldwide, but sensitivity for CRC ranges between 53%-99% depending on the cut-off values used, whereas sensitivity for advanced adenomas is disturbingly low (39%-57%).

The aim of this study is to evaluate the diagnostic accuracy of the AeonoseTM to distuinguish people with CRC from healthy controls.

DETAILED DESCRIPTION:
Rationale: An electronic nose (eNose) is an artificial olfactory system that analyses volate organic compounds (VOCs) in exhaled breath. Exhaled human breath is mainly composed of inorganic compounds, inert gases and VOCs. VOCs are exhaled in very low concentrations and reflect pathological processes such as inflammation, oxidation, infection and neoplasms. The perspective is that metabolic and biochemical processes in several pathological situations cause different endogenous VOCs to arise, were they can serve as non-invasive biomarkers for certain diseases.

Primary objective: To evaluate the diagnostic accuracy of the AeonoseTM to distinguish the breathing pattern from patients with colorectal cancer from healthy controls using the previously established breathing pattern.

Secondary objecitves:

* To evaluate the diagnostic accuracy of the AeonoseTM to distinguish the breathing pattern from patients with polyps (e.g. advanced adenomas, sessile serrated lesions).
* To determine the influence of colonic cleansing (laxative use) on breathing patterns.

Study population: Adult patients referred for colonoscopy.

Estimated sample size: 66 patients with CRC.

Intervention: Participants will be asked to breath through the AeonoseTM for 5 minutes. There are no risks, nor benefits for the participants.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Suspicion for (pre-)malignant lesions of the colon scheduled for colonoscopy

Exclusion Criteria:

* Subjects with other known malignancies
* Subjects with established inflammatory bowel disease

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
sensitivity/specificity for CRC | 38 weeks
  Diagnostic accuracy of the Aeonose to detect CRC in terms of sensitivity and specificity

SECONDARY OUTCOMES:
sensitivity/specificity for advanced adenomas and/or sessile serrated lesions. | 38 weeks
  Diagnostic accuracy of the Aeonose to detect polyps in terms of sensitivity and specificity
Sensitivity/specificity for detection of CRC and/or polyps before and after bowel preparation | 38 weeks
  Diagnostic accuracy, sensitivity/specificity/AUC

CONTACTS AND LOCATIONS:
Locations (1):
- Medisch spectrum Twente, Enschede, Twente, Netherlands

REFERENCES:
- [Derived] van Keulen KE, Jansen ME, Schrauwen RWM, Kolkman JJ, Siersema PD. Volatile organic compounds in breath can serve as a non-invasive diagnostic biomarker for the detection of advanced adenomas and colorectal cancer. Aliment Pharmacol Ther. 2020 Feb;51(3):334-346. doi: 10.1111/apt.15622. Epub 2019 Dec 20. PMID 31858615